CLINICAL TRIAL: NCT04618653
Title: Development of a Comprehensive and Dynamic AA Process Model: One Day at a Time
Brief Title: Comprehensive Process Model of AA-related Behavior Change
Status: Active, not recruiting | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Scott Tonigan, CASAA Director, University of New Mexico
Other Study IDs: 1525759-3
Record Dates: First submitted 2020-10-16; First posted 2020-11-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early AA Attenders with Alcohol Use Disorder: observational study that includes three fixed assessments (Baseline, 3, and 6-month). Subset of participants will also provide daily EMA data.
  Interventions: Other: assessment only

INTERVENTIONS:
Other: assessment only — Three assessment will include computerized assessments, interviews, and subset will provide daily reports of prescribed AA behaviors and practices

SUMMARY:
Alcoholics Anonymous (AA) is one of the most popular resources for dealing with alcohol-related problems, and 12-step therapy (TS), based upon AA doctrine and practice, is one of the prevailing alcohol treatment approaches in the United States. Two large multisite trials, one high in internal validity and the second high in external validity came to the same conclusion, TS was equally effective as more research supported therapies, and may actually be superior when total abstinence is the treatment goal. A primary objective of TS is to facilitate AA affiliation and strong evidence suggests that this aim is a major factor accounting for the effectiveness of TS. High priority has therefore been assigned to the investigation of what actually occurs in AA, with a special focus on identifying prescribed AA behaviors and processes that are predictive of drinking reduction. The guiding assumption of these efforts is that the key to improve TS is to first understand AA better. To this end, this study will generate, for the first time, a comprehensive and definitive process model of AA-related behavior change. This objective will be realized through the highly innovative use of EMA data collection among early AA affiliates. Using real-time daily data, aim 1 will determine if four MOBC identified by AA researchers (gains in social support, increased abstinence self-efficacy, spiritual practices, and negative urgency) mediate the linkage between three types of AA prescribed behaviors and drinking outcome. Noteworthy, these analyses will include the first rigorous testing of six of seven of criteria to confirm (or reject) that these four statistical mediators are MOBC. Aim 2 will investigate whether the actions of the AA active ingredients on mediators (a path) and the actions of the mediators (b path) are constant over time or, alternatively, if there are critical periods of influence. Last, aim 3 will determine if the four MOBC operate differently across distinct subpopulations. To achieve study aims, we propose a two-group randomized longitudinal study (N = 190). In one group (n = 130) we will collect 6-months of continuous EMA data, allowing us to examine near real-time associations between AA active ingredients in three domains, four MOBC, and drinking. In tandem, we will also conduct in-person interviews at baseline, 3, and 6-months. Assessment reactivity is a concern, especially so because this will be the first study to use EMA in addition to in-person interviews in AA research. We will therefore include a traditional fixed assessment group (n = 60) also interviewed at baseline, 3, and 6-months to identify potential measurement biases introduced in our innovative approach. Achievement of study aims will generate the first empirically validated AA process model that will inform TS with critical information for improving treatment outcomes.

DETAILED DESCRIPTION:
Recruitment. Adults will be recruited at AA clubs and other AA meeting locations in Albuquerque, NM. We have previously recruited from these AA clubs and have a solid record of achieving our recruitment goals. We will recruit and consent 4 participants per month. Recruitment efforts will begin in month 3 (year 01) and will continue until month 49 (year 4). Recruitment will be unrestricted with regard to gender and minorities. We expect that racial/ethnic diversity will be consistent with our past AA studies with similar inclusion/exclusion criteria (54-65% male, 41-43% Hispanic. Based on considerable expertise, research staff will recruit participants from AA club lounge areas (which will result with the staff member providing a study advertisement flyer to the prospect) or directly through flyers posted in AA clubs (detailed background information provided). Interested prospects will first complete a stage 1 eligibility screen via a web-based application (link provided on flyer) or through a telephone interview with research staff (phone number provided on flyer). All inclusion/exclusion criteria will be collected in stage 1 screening with the exceptions of inclusion criterion #1 (ADS) and exclusion criterion #4 (active psychosis/in ability to provide documented informed consent). Prospects that are deemed eligible and who remain interested will have an appointment scheduled at CASAA for stage 2 screening. In addition to verifying stage1 screening information, in stage 2 our research staff will administrer the ADS and determine if the prospect is actively psychotic and capable (or not) to provide informed consent.

Randomization/Consent. After stage two screening, eligible clients who remain interested will be told the following by research staff, "It looks like this study is a good fit for you. The study has two groups, one involves a little time each day for six-months and it requires three in-person interviews, one today, the second in three-months, and then a six-month interview. The second group requires less time and effort on your part and, as a result, does not offer as much compensation. This second group has only three interviews, one today, the second in three-months, and then a six-month interview. Assignment to one of these groups is entirely random. To help you decide if you want to participate in this study we can tell you that you have about a one in three chance of being assigned to the low-effort compensation group. Do you have any questions? If not, would you like to participate this study?" Eligible prospects willing to proceed will then be randomized using the urn procedure. Urn variables are: (1) total ADS score, (2) PDA (past 90 days), and (3) percent days of AA attendance (past 90 days). Using data from two prior AA studies with similar inclusion/exclusion criteria, we calculated the median for these three variables. Our high-low values for this study are: AA attendance (8 or fewer days = 1, 9 or more days = 2), ADS (0-47 = 1, 48 and higher = 2), and PDA (0 to .55 = 1 and .56 to 1.0 = 2). Once group assignment has been determined, the RA will initiate the consent process with the consent form that corresponds to the assigned group. Participants electing to provide consent will be administered a breathalyzer test prior to signing of informed consent (must have a blood alcohol level < .05 to be consented). A consented person who has not completed the baseline assessment after two weeks of consenting date will be regarded as inactive and their "slot" in the study will be filled with another person. We have discussed and developed this consenting procedure in collaboration with the UNM IRB staff

In-Person Assessments. All study participants will be interviewed and complete self-report questionnaires at baseline, 3, and 6-months. These battery's (Table 2; Appendix A), have 3 semi-structured interviews and 9 self-report questionnaires. All assessments have strong psychometric properties and will be administered by trained project research staff in an office dedicated to research assessment. To reduce the influence of assessment order effects, self-report questionnaires will be rotated, and the order of self-report and semi-structured interviews will also be rotated across assessment points.

Table 2. Proposed In-Person Assessment Battery Assessment Type of Assessment Intake 3-mo 6-mo Screening Form (stage 1 and 2) Structured Interview X Informed Consent Structured Interview X Locator Form Structured Interview X p.r.n. p.r.n. Demographic Interview Structured Interview X Alcohol Dependence Severity (ADS) Self-Report X Form 90 - (Healthcare/Substance Use) Structured Interview X X X Drinker Inventory of Consequences (DrInC) Self-Report X X X Twelve-Step Participation Questionnaire (TSPQ) Self-Report X X X Important People and Activities (IPA) Structured Interview X X X Group Environment Scale (GES) Self-Report X X X What I got From Treatment (WFT) Self-Report X X X General AA Tools of Recover (GAATOR) Self-Report X X X Religious Practices and Beliefs (RPB) Self-Report X X X Alcohol Abstinence Self-Efficacy Scale (AASE) Self-Report X X X UPPS Impulsive Behavior Scale Self-Report X X X

D.8.b. Scheduling Follow-up Interviews. At the end of the baseline assessment, research staff will schedule a date for the 3-month follow-up interview with each participant (N = 190). At this time, locator and contact information will be reviewed for accuracy. About 2 weeks before the scheduled 3-month interview, we will initiate a reminder using phone and/or mail, as necessary. All participants will have access to public transportation fare, if needed. At the end of the 3-month interview research staff will schedule the 6-month interview, review contact information with the participant, and repeat the two-week reminder call. Regardless of whether or not a 3-month interview had been conducted every possible effort will be made to locate, schedule, and conduct the 6-month interview. All 3 and 6-month interviews will be conducted at CASAA.

D.8.c. Follow-Up Procedures and Attrition. Our research staff specializes in follow-up tracking of clinical samples. Specifically, our staff is highly experienced in using state-of-the-art techniques in locating and scheduling clients for interviews, e.g., multiple locator information, postal system, MVD checks, reverse phone directories, house calls, internet credit searches, county, state, and national death registries. All our procedures are IRB approved, and are explained to prospective study participants before obtaining informed consent. We are confident that we can achieve an 80-85%% follow-up rate at the three and six-month follow-up. Explained, when we conducted a 10-year follow-up of the Project MATCH outpatient sample recruited in Albuquerque, seven years had elapsed without participant contact of any kind. Of the 181 surviving participants that consented for a long-term follow-up at the 3-year interview (22 had died) we successfully interviewed 148 (82%).

ELIGIBILITY:
Inclusion criteria:

1. ADS score ≥ 8 (past 12 months)
2. alcohol use, past 4 months
3. attended ≥ 1 AA meeting, past three months
4. ≥ 18 years of age
5. speak and read English at the sixth grade level.

Exclusion Criteria:

1. ≥ 4 months of continuous AA attendance (lifetime), with continuous defined as attending at least 1 AA meeting per week over a 4-month period
2. admitted into inpatient or outpatient substance abuse treatment in the prior 12 months (currently seeking treatment will not be a basis to exclude)
3. unable to provide the names of two locators
4. active psychosis or a condition impairing ability to provide informed consent
5. pending legal convictions involving ≥ 90-days incarceration
6. plans to relocate to another state
7. ≥ 3 formal treatment experiences (lifetime) for substance abuse
8. ≥ 12 months of continuous abstinence from alcohol (lifetime) initiated in response to perceived alcohol-related problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Percent abstinent days at baseline, 3 months and six-months | baseline, 3, and 6, months
  calculated as the number of abstinent days in an assessment window divided by the total number of days in an assessment window
Change in daily Percent abstinent days baseline to six-months | baseline to six-months
  mobile device will provide daily reported drinking

CONTACTS AND LOCATIONS:
Overall Officials: JEFFREY TONIGAN, phd, Principal Investigator — UNIVERSITY OF NEW MEXICO (CASAA); Matthew r Pearson, phd, Study Director — UNIVERSITY OF NEW MEXICO (CASAA)
Locations (1):
- Center on Alcohol, Substance Use, and Addictions (CASAA), Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No